CLINICAL TRIAL: NCT01930643
Title: Effect of Electric Muscle Stimulation on Patients With Chronic Respiratory Failure
Brief Title: Electric Muscle Stimulation for Patients With Chronic Respiratory Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment and change of faculty
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Kuang-Hua Cheng, MD, Visiting staff, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13MMHIS070
Record Dates: First submitted 2013-08-25; First posted 2013-08-29 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Chronic Respiratory Failure; Critical Illness Myopathy
Keywords: Electric muscle stimulation; mechanical ventilation; chronic respiratory failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electric muscle stimulation(EMS) (Experimental): EMS:use programmed middle frequency electric stimulation device(HELEX 573)for both quadriceps stimulation, 32 minutes per day, 5 time per week.
  Interventions: Device: EMS
- Control (No Intervention): Patients with routine passive rehabilitation program.

INTERVENTIONS:
Device: EMS — HELEX 573 : strength aggravation mode with middle frequency carrier(1500Hz), minimal voltage for visible muscle contraction(maximum output is 75mA) , 32 minutes per day.
  Arms: Electric muscle stimulation(EMS)

SUMMARY:
Background: After mechanical ventilation, 5-20% of patients with acute respiratory failure would depend on ventilator support more than 14 days because of critical-illness weakness and their underlying diseases such as heart failure and chronic obstructive pulmonary disease.

Hypothesis: Electric muscle stimulation(EMS) will improve their muscle strength and shorten their ventilator days.

Design: Randomized controlled trial. Adult patients with mechanical ventilation more than 14 days are eligible. EMS would be applied in experimental group 32 minutes/day on their bilateral thigh.

DETAILED DESCRIPTION:
Randomized controlled trial involves the adult patients with invasive mechanical ventilation more than 14 days. The participants were not eligible for active rehabilitation because of drowisness or weakness(Medical Research Council (MRC) Scale for Muscle Strength≦ Grade 3).

EMS would be applied in experimental group 32 minutes/day on their bilateral thigh(quadriceps muscle).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient required mechanical ventilation more than 14 days
* No ability for active endurance exercise because of poor consciousness or limb weakness.

Exclusion Criteria:

* Pregnant women
* Limb wound/infection interfered with electric pad application
* Recent acute myocardial infarction or life-threatening arrhythmia
* Uncontrolled epilepsy
* Dying patients without attempt of ventilator weaning
* Absence of respiratory drive

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08-21 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuang H Cheng, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electric Muscle Stimulation(EMS) | Control
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electric Muscle Stimulation(EMS) | Control | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 6 | 5 | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 82 [74 to 83] | 73.5 [66 to 75] | 75 [73 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  Taiwan | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Ventilator-free Days
Description: the cumulative ventilator-free days after intervention, in following 28 days.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Electric Muscle Stimulation(EMS) | Control
Number analyzed (Participants) | 7 | 6
day | 6 [0 to 17] | 0 [0 to 19]

2. Secondary Outcome: Grip Power
Description: Weekly improvement of both hand grip muscle power in kilogram(Kg)
Time Frame: 7 days after intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The first 14 days after Electric Muscle Stimulation is applied
Arm/Group | Electric Muscle Stimulation(EMS) | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes